CLINICAL TRIAL: NCT06791720
Title: Effects of Music-with-Movement (Simultaneous Cognitive-motor Dual-task Training) on Cognitive and Physical Performance of People With Potentially Reversible Cognitive Frailty: a Randomised Controlled Trial
Brief Title: Effects of Music-with-Movement on Cognitive and Physical Performance of People With Potentially Reversible Cognitive Frailty: a Randomised Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Deakin University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20241202003
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Physical Frailty; Mild Cognitive Impairment (MCI); Cognitive Frailty
Keywords: Music-with-Movement; Cognitive-Motor; Dual-Task; Physical Performance; Cognitive Performance; Cogntive Frailty; Intervention
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A single-blinded, two-arm randomized controlled trial will be adopted to evaluate the effects of the Music-with-Movement Simultaneous Cognitive-Motor Dual-Task Training (MM-SDTT) on the cognitive and physical performance of older adults with cognitive frailty. Participants will be randomized to either the treatment or social control groups at a 1:1 ratio using permuted block randomization with a block size of 2.
Who Masked: Outcomes Assessor
Masking Description: The researchers who perform the outcome assessment and analysis will be blinded to the group allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music-with-Movement Simultaneous Cognitive-Motor Dual-Task Training (MM-SDTT) group (Experimental): Participants in the treatment group will undergo a 16-week MM-SDTT program, which includes once-weekly center-based sessions and twice-weekly home-based sessions. Center-based sessions will be supervised by an interventionist with a physical fitness background, while participants will have home-based sessions using provided training videos.
  Interventions: Behavioral: music-based cognitive-motor dual-task training/exercise
- Social Control Group (Other): Participants in the social control group will have social chatting weekly for 45 minutes over 16 weeks, to control the potential social effect of the MM-SDTT on cognitive functions. Remedial MM-SDTT will be delivered to the social control group after the data collection is completed.
  Interventions: Behavioral: Social Gatherings

INTERVENTIONS:
Behavioral: music-based cognitive-motor dual-task training/exercise — Participants is engaged in 4 sessions for each training, including rhythmic marching, singing familiar songs, dance workout with elastic bands and stretching exercise with relaxing music. This combination of physical and cognitive activities aims to improve overall well-being by integrating music and movement, making the exercise both enjoyable and beneficial for mental and physical health. Rhythmic aerobic exercises to music focuses on rhythm and movement accuracy. Listening and singing familiar songs is cognitively stimulating. Dance workout allows strength and endurance training with music. Stretching exercise with relaxing music improves the range of movement in major muscle and tendon groups.
  Arms: Music-with-Movement Simultaneous Cognitive-Motor Dual-Task Training (MM-SDTT) group
Behavioral: Social Gatherings — Participants in the social control group will have a social gathering at the participating center once weekly over the 16 weeks. They will also continue to receive the usual care offered by the centers, such as social support, and health education.
  Arms: Social Control Group

SUMMARY:
This study aims to evaluate the effects of Music-with-Movement Simultaneous Cognitive-Motor Dual-Task Training (MM-SDTT) on cognitive and physical performance in older adults with cognitive frailty coexisting with mild cognitive impairment (MCI) and physical frailty.

Research Questions:

1. Will the treatment group show greater improvement in global cognitive functions than the social control group at Week 16?
2. Will the treatment group show greater improvements in both cognitive, physical performance and psychosocial well-being than the social control group at Weeks 16 and 28?

Methodology:

Participants in the Treatment Group:

* Undergo a 16-week intervention comprising:

  1. Once-weekly center-based training supervised by a physical coach
  2. Twice-weekly home-based training using provided training videos

     Participants in the Social Control Group:
* Engage in once-weekly social gatherings and receive remedial training after data collection is completed.

DETAILED DESCRIPTION:
There is a need to enhance the well-being of older adults with cognitive frailty, defined as the coexistence of mild cognitive impairment (MCI) and physical frailty. Literature shows that combining physical training with cognitive training is effective to improve the health outcomes of MCI, while whether it is beneficial to those MCI with co-existing physical frailty is unknown.

The proposed 16-week Music-with-Movement Simultaneous Cognitive-Motor Dual-Task Training (MM-SDTT) aims to evaluate its effects on the cognitive and physical performance of older adults with cognitive frailty. The MM-SDTT is designed to engage participants through music with cognitive and physical training. The intervention will include warm-up exercise, rhythmic marching, singing familiar songs, dancing workout, stretching exercise with relaxing music, and cool-down exercise. The intervention protocol has been designed according to the guidelines of the American College of Sports Medicine and evidence of previous music-with-movement intervention research.

The study will recruit older adults aged 60 and above, who live in the community and can walk independently, and also have cognitive frailty. Participants will be randomly assigned to either the treatment group or a social control group. Participants in the treatment group will undergo 16-week MM-SDTT consisting of once-weekly center-based training supervised by a coach and twice-weekly home-based training with provided training videos. The logbook and wearable sensor will be used as tools to monitor and record physical activity. Participants in the social control group will participate in social gatherings once weekly over the 16 weeks without affecting the usual care. The MM-SDTT is expected to improve the cognitive and physical functions of older adults with cognitive frailty.

The protocol aims to evaluate the immediate effects (sixteen weeks after weekly supervised sessions, i.e. on the 16th week) and the mid-term effects (three months when the intervention has been completed, i.e. on the 28th week). Hypotheses include that the treatment group will show greater improvements in global cognitive functions compared to the control group at Week 16, as well as greater enhancements in physical and cognitive performance than the control group at Week 16 and 28.

Overall, this research addresses the research gap in interventions for older adults with cognitive frailty, aiming to provide an evidence-based approach to improve their cognitive and physical health outcomes. The anticipated findings might have significant implications for the development of early-stage interventions and clinical practice that can enhance the quality of life for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 and above;
* Community-dwelling, as defined by living at home and not having stayed in a long-term care facility in the last 12 months as reported by the participants;
* Able to walk independently or with a stick;
* A cutoff value of = 0 in the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) indicates the participants' physical stability;
* A cutoff score of = 0.5 in the Clinical Dementia Rating indicates participants with Mild Cognitive Impairment (MCI);
* A cutoff score of ≥1 on the FRAIL Scale indicates participants with physical frailty;

Exclusion Criteria:

* Is suffering from any critical medical or psychiatric illness;
* Has an uncorrectable visual and/or hearing impairment that hinders the participation;
* Is having the MCI or physical frailty only;
* Is participating in other trials;
* Chronic use of corticosteroids, immunosuppressive drugs, androgen-, estrogen-, or progestin-containing compounds
* Taking psychotropic, antiarrhythmic, or hypnotic medications
* Advised by healthcare professionals (e.g., physicians or physiotherapists) not to participate in moderate-to-vigorous exercises.
* Older adults with special conditions or increased risk of injuries that require substantial adjustment in exercise regime, including those with COPD, renal disease, cancer, etc.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | Change from baseline to 28 weeks after programme
  The Montreal Cognitive Assessment (MoCA) is a test of global cognitive functions. MoCA consists of 8 domains, including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The scores range from 0 to 30, with higher scores indicating better cognitive functions.

SECONDARY OUTCOMES:
Frontal Assessment Battery | Change from baseline to 28 weeks after programme
  The Frontal Assessment Battery (FAB) is a test of executive functions. It consists of 6 domains, including conceptualization, mental flexibility, programming, sensitivity to interference, inhibitory control, and environmental autonomy, on a 3-point numeric scale. The scores range from 0 to 18 points, with a higher score indicating better executive functioning.
Fuld Object Memory Evaluation | Change from baseline to 28 weeks after programme
  The Fuld Object Memory Evaluation (FOME) is a test of memory functions, such as encoding, storage, recalling across five trials, and a delayed recall trial. There are three FOME scores, which include total storage (range from 0-50), total retrieval (range from 0-50), and delayed recall (range from 0-10). Higher total scores refer to better memory functions.
Modified Fuld Verbal Fluency Test | Change from baseline to 28 weeks after programme
  The Modified Fuld Verbal Fluency Test (MFVT) is used to test verbal fluency, which is embedded in the FOME as a distraction task. Total scores are the total number of items being named, with higher scores indicating better verbal fluency.
Social Participation Quesionnaire | Change from baseline to 28 weeks after programme
  The Social Participation Questionnaire (SPQ) is used to test the level of social participation. It consists of 17 questions including informal social contact, social contact through activities in public spaces, participation in group activities, and participation in community groups, on a 6-point numeric scale from 0 to 5. The scores range from 0 to 85 points, with higher scores indicating better social participation.
Subjective Happiness Scale | Change from baseline to 28 weeks after programme
  The Subjective Happiness Scale (SHS) is a 4-item scale of global subjective happiness. Each item is rated on a 7-point Likert scale from 1 to 7, and item #4 is reverse coded. All item scores are averaged to get the total scores which range from 1 to 7 with a higher score indicating greater happiness.
DeJong Gierveld Loneliness Scale | Change from baseline to 28 weeks after programme
  The DeJong Gierveld Loneliness Scale (DJGLS) is a 6-item scale of emotional loneliness and social loneliness. On the negatively worded items 1-3, the score of Yes = 1, More or less = 1, and No = 0. On the positively worded items 4-6, the score of Yes = 0, More or less = 1, and No = 1. All item scores are averaged to get the total scores which range from 1 to 6 with a higher score indicating greater loneliness.
Edmonton Frail Scale | Change from baseline to 28 weeks after programme
  The Edmonton Frail Scale (EFS) is a test to measure frailty. It consists of 9 questions with multidimensional aspects of frailty, including cognition, general health status, functional independence, social support, medication use, nutrition, mood, and continence. The scores range from 0 to 17, with higher scores indicating more severe frailty.
Timed Up and Go Test | Change from baseline to 28 weeks after programme
  The Timed Up and Go Test (TUG) is a test of physical functional abilities. A shorter duration of completing the test indicates better mobility.
Handgrip Strength | Change from baseline to 28 weeks after programme
  Handgrip strength is measured with a hand dynamometer to indicate muscle strength.
Six-minute Walk Test | Change from baseline to 28 weeks after programme
  The Six-Minute Walk Test (6MWT) measures aerobic fitness and endurance by assessing the distance a participant can walk in six minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Justina Liu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For confidentiality, the data will be kept anonymous and the information of all participants will be replaced by reference codes. The data will be kept in a locked place and electronic versions will be encrypted, and only be accessible by the researchers. All data will be destroyed within 7 years after the completion of this research.

REFERENCES:
- [Background] Liu JYW, Kwan RYC, Yin YH, Lee PH, Siu JY, Bai X. Enhancing the Physical Activity Levels of Frail Older Adults with a Wearable Activity Tracker-Based Exercise Intervention: A Pilot Cluster Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Sep 30;18(19):10344. doi: 10.3390/ijerph181910344. PMID 34639644
- [Background] Kwan RY, Lee D, Lee PH, Tse M, Cheung DS, Thiamwong L, Choi KS. Effects of an mHealth Brisk Walking Intervention on Increasing Physical Activity in Older People With Cognitive Frailty: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 31;8(7):e16596. doi: 10.2196/16596. PMID 32735218
- [Background] Cheung, D.S.K., et al., Music-with-movement intervention for people with mild/early cognitive impairment: An effectiveness-implementation hybrid cluster randomized controlled trial. Alzheimer's & dementia, 2020. 16: p. n/a.
- [Background] Cheung DSK, Lai CKY, Wong FKY, Leung MCP. Is music-with-movement intervention better than music listening and social activities in alleviating agitation of people with moderate dementia? A randomized controlled trial. Dementia (London). 2020 Jul;19(5):1413-1425. doi: 10.1177/1471301218800195. Epub 2018 Sep 20. PMID 30235949
- [Background] Cheung DSK, Lai CKY, Wong FKY, Leung MCP. The effects of the music-with-movement intervention on the cognitive functions of people with moderate dementia: a randomized controlled trial. Aging Ment Health. 2018 Mar;22(3):306-315. doi: 10.1080/13607863.2016.1251571. Epub 2016 Nov 7. PMID 27819483
- [Background] Chen YL, Pei YC. Musical dual-task training in patients with mild-to-moderate dementia: a randomized controlled trial. Neuropsychiatr Dis Treat. 2018 May 30;14:1381-1393. doi: 10.2147/NDT.S159174. eCollection 2018. PMID 29881275
- [Background] Tait JL, Duckham RL, Milte CM, Main LC, Daly RM. Influence of Sequential vs. Simultaneous Dual-Task Exercise Training on Cognitive Function in Older Adults. Front Aging Neurosci. 2017 Nov 7;9:368. doi: 10.3389/fnagi.2017.00368. eCollection 2017. PMID 29163146
- [Background] Satoh M, Ogawa J, Tokita T, Nakaguchi N, Nakao K, Kida H, Tomimoto H. The effects of physical exercise with music on cognitive function of elderly people: Mihama-Kiho project. PLoS One. 2014 Apr 25;9(4):e95230. doi: 10.1371/journal.pone.0095230. eCollection 2014. PMID 24769624
- [Background] Murrock CJ, Higgins PA. The theory of music, mood and movement to improve health outcomes. J Adv Nurs. 2009 Oct;65(10):2249-57. doi: 10.1111/j.1365-2648.2009.05108.x. PMID 20568327
- [Background] Sarkamo T. Cognitive, emotional, and neural benefits of musical leisure activities in aging and neurological rehabilitation: A critical review. Ann Phys Rehabil Med. 2018 Nov;61(6):414-418. doi: 10.1016/j.rehab.2017.03.006. Epub 2017 Apr 29. PMID 28461128
- [Background] Tam ACY, Chan AWY, Cheung DSK, Ho LYW, Tang ASK, Christensen M, Tse MMY, Kwan RYC. The effects of interventions to enhance cognitive and physical functions in older people with cognitive frailty: a systematic review and meta-analysis. Eur Rev Aging Phys Act. 2022 Aug 24;19(1):19. doi: 10.1186/s11556-022-00299-9. PMID 36002799